CLINICAL TRIAL: NCT03882671
Title: Development of a Minimally Invasive Seizure Gauge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seer Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HREC042_18
Record Dates: First submitted 2019-03-11; First posted 2019-03-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Monitoring Device (Experimental): Subjects will be asked to wear up to 3 different noninvasive seizure detection devices including EpiTel EpiLog, Empatica E4, GeneActiv
  Interventions: Device: EpiTel Epilog; Device: Empatica E4; Device: GENEActiv

INTERVENTIONS:
Device: EpiTel Epilog — EEG recording device
Device: Empatica E4 — PPG, sweat level, temperature and accelerometry recording device
Device: GENEActiv — Temperature, light level and accelerometry recording device

SUMMARY:
The researchers are trying to assess changes in physiological signals before and during seizures.

DETAILED DESCRIPTION:
Subjects that are undergoing video EEG monitoring in their home for their epilepsy at Seer Medical will be consented to participate in this study for a minimum of two days and/or the duration of their monitoring period for their clinical care. Subjects will be asked to wear up to 4 different commercially available seizure detection devices and complete surveys.

When the subjects clinical EEG monitoring is completed data scientists will analyze the data to identify patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy undergoing scalp EEG for clinical care, or an implanted device capable of monitoring brain activity and identifying seizures
* Patients of age 18 or above

Exclusion Criteria:

* Cognitive or psychiatric condition rendering patient unable to cooperate with data collection, or manage and recharge smart watch and tablet computer devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Multimodal Assessment of Physiological Signals During Seizure Events Measurable with Wearable Sensors | 2-7 days approximately
  We will collect physiological signals with the three wearable, noninvasive biosensors in Seer Medical patients undergoing scalp-recorded video EEG-ECG as part of their clinical epilepsy evaluation. These signals include temperature, light level, EEG, heart rate, galvanic skin response, PPG, accelerometry. We will evaluate biosignals based on reliability to detect seizures.
Wearable Sensors Comfort Assessment | 2-7 days approximately
  We will collect physiological signals with the three wearable, noninvasive biosensors in Seer Medical patients. We will evaluate subject comfort and ease of use for each device, measured through quantitative surveys.
Seizure Detection and Prediction using Multimodal Physiological Data | 2-7 days approximately
  We will apply data mining and machine learning methods to identify patterns in the collected physiological signals and correlate these patterns with the timing of seizures identified by the patient's clinical video-EEG monitoring. We will use sensitivity and specificity measures to determine which signals are most useful in detecting and predicting seizure events.

CONTACTS AND LOCATIONS:
Overall Officials: Dean R Freestone, PhD BEng, Principal Investigator — CEO
Locations (1):
- Seer Medical, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No